CLINICAL TRIAL: NCT05562869
Title: Belatacept as a Replacement for CNIs 3 to 12 Months Post-transplantation in Patients With Early Graft Dysfunction
Acronym: BELASBRIDGE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC21_0587
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Chronic Kidney Failure
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: transient belatacept (Experimental): IV, 5mg/Kg days 1, 15, 30, 45 and 60 then every months
  Interventions: Drug: Belatacept 250 Milligram Intravenous Powder for Solution

INTERVENTIONS:
Drug: Belatacept 250 Milligram Intravenous Powder for Solution — Phase 1 (from 3 to 12 months post transplantation): conversion to belatacept (IV, 5mg/Kg days 1, 15,30, 45, 60 then every months) and CNI withdrawal.
  Phase 2 (from 12 to 18 months post transplantation) : belatacept arrest and CNI resumption (tacrolimus target 6 ng/ml)

SUMMARY:
Calcineurin inhibitors (CNI) remain the standard treatment in renal transplantation to prevent rejection. Currently the main limitation of kidney transplantation is the occurrence of chronic graft dysfunction due to the CNI nephrotoxicity. Thus, strategies to minimize or stop CNI have been developed as belatacept, a fusion protein (CTLA4-Ig) blocking the ligand of the main CD28 costimulatory molecule. In the original phase III trial, used de novo in combination with MMF (without CNI) belatacept allowed to obtain a better renal function as soon as 1 year and a better graft and patient survival after 7 years. Despite these excellent results, belatacept has not become the gold standard due to a higher incidence of early rejection. In addition, belatacept is not covered by the french social security policy, because benefits are considered insufficient with respect to the cost. Patients with poor early graft function are a preferred indication of belatacept. It is then used instead of CNI at 3 months post-transplant allowing to improve kidney function without over-risk of rejection. Currently after conversion, belatacept is maintained indefinitely due to the supposed CNI chronic nephrotoxicity. However this one is more and more questionable. Thus, the investigators assume that in patients with poor function at 3 months posttransplantation the belatacept's benefit could be obtained by a transient replacement of CNI by belatacept from 3 to 12 months post-transplantation. It is the feasibility of this strategy and its medico-economic impact that the investigators wish to study.

DETAILED DESCRIPTION:
The standard maintenance regimen in renal transplantation combines calcineurin inhibitor (CNI: ciclosporin or tacrolimus) and anti-metabolite drugs (mycophenolate mofetil (MMF) or mycophenolic acid (MPA)). CNI in the 1980s made kidney transplantation possible by drastically reducing acute rejection rates in the first year. Currently the main limitation of kidney transplantation is the occurrence of chronic graft dysfunction. While half of patients die with a functional graft, the other half return to dialysis and require retransplantation. Paradoxically, CNI has been identified as a leading cause of chronic graft dysfunction. Indeed, these molecules are nephrotoxic both : acutely and transitory due to a vasoconstrictor effect that modulates intra-renal hemodynamic and chronically due to extensive fibrosis. In the late 1990s, with the development of a new class of immunosuppressants, mammilian target of rapamycin (mTor) inhibitors (sirolimus and everolimus), CNI-free protocols were developed. The results were disappointing due in part to the undesirable effects of these treatments and secondly to the occurence of chronic rejections related to the appearance of Donor Specific Antibody (DSA) antibodies.

Finally in the mid-2000s belatacept is a fusion protein (CTLA4-Ig) blocking the ligands of the main costimulatory molecule (CD28) emerged. In the Phase III princeps assay (BENEFIT), this molecule was used as a maintenance treatment following transplantation (de novo) in combination with MMF (without CNI). Compared to the control group with CNI, patients receiving belatacept had better renal function from 1 year and after 7 years survival (graft and patient) were better. These benefits were attributed, on the one hand, to the absence of CNI and, on the other hand, to a very good control of the alloimmune response demonstrated by a lower incidence of DSA in the belatacept group.

Despite these excellent results, belatacept has not become the gold standard in renal transplantation for two main reasons. First, when it is used de novo (as in BENEFIT), there is a significant incidence of early rejection, known as "costimulation blockade resistant". The second issue is medico-economic. Indeed, to date and despite the accumulation of favorable data, in France and in most countries, belatacept has marketing authorization but is not supported by social security policy due to benefits regarded as insufficient with respect to the cost (related to the IV administration requiring hospital environment every month).

Consequently, it is important to precise which recipients may benefit more from this molecule. Patients, often elderly, with poor early function of the graft due to the poor quality of a marginal / "extended criteria" donor, are a good indication of belatacept not used de novo but after 3 months instead of CNI. This conversion most often allows to significantly improve the renal function of these patients to a much more acceptable level which remains stable beyond and without cost in terms of rejection (probably because of the time interval with the transplant). In this situation, several series reported success rates ranging from 80 to 100% with a rejection incidence between 0 and 20%. Failures are most often due to patients with non-primary graft function.

Currently after the conversion, belatacept is always maintained indefinitely most often in association with MMF. This usage generates significant costs and in fact, limits the access of belatacept for other patients. This practice is based on the dominant idea that chronic nephrotoxicity of CNI is the cause of chronic graft dysfunction.

However, while reversible acute toxicity, mediated by hemodynamic changes in intra-renal vascularization, is undeniable, the importance and even the reality of chronic, cumulative, irreversible CNI toxicity has been questioned during the last decade, while the importance of chronic anti-donor antibody (DSA) rejection to explain chronic graft dysfunction was demonstrated. The chronic toxicity of CNI is probable when high doses are necessary to prevent rejection during the first year but uncertain beyond.

Thus, the investigators assume that in patients with poor graft function at 3 months post-transplantation most of the benefit of belatacept could be obtained by a transient replacement of CNI from 3 to 12 months post-transplantation.

Indeed, in these often elderly patients, who have most often received an "extended criteria" graft (derived from a marginal donor), presenting chronic lesions, CNI-induced intra-renal vasoconstriction could more easily evolve to irreversible lesions in the context of ischemia-reperfusion inherent in the graft itself. At 1 year after transplantation the reintroduction of CNIs at minimized doses could only moderately alter the renal function allowing to maintain them at long term.

The purpose of this study is to demonstrate the feasibility of this transient treatment strategy (from 3 to 12 months post transplantation) in patients with poor function at 3 months.

From 3 months post-transplantation, patients will receive for 9 months (phase 1) a treatment with belatacept allowing to stop CNI. Then CNI will be reintroduced (phase 2) with a follow-up period of 6 months which will make it possible to judge the feasibility of this strategy.

Belatacept is the only biotherapy introduced successfully in transplantation. But this treatment, because of the limitations raised, has not yet found a definite place. Our project is to study a practical question: can the investigators stop belatacept after having introduced it early in the context of an early dysfunction while preserving the benefits. The decisive contribution of this study would be to prove the concept of a transient treatment by belatacept which has not been reported. The medico-economic consequences would be major, the cost of a long-term treatment by belatacept, especially because of its administration in hospital, being much higher than that of a conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* adult older than 18 years old.
* transplantation of a deceased or living donor kidney (non-human leukocyte antigen(HLA)-identical) with blood type (ABO) compatibility
* no contraindication to the protocol graft biopsy (10 weeks post transplant)
* treatment by CNI / MPA +/- prednisone
* renal function estimated by creatinine clearance according to CKD-EPI <30 ml / min / 1.73m2.
* having no difficulty in understanding and communicating with the investigator and his representatives.
* Agreeing to give informed written consent
* benefiting from a Social Security policy.
* results of the 10-week post-transplant renal biopsy finding no rejection or BK virus (member of the polyomavirus family) nephropathy, no recurrence, no thrombotic microangiopathy, no cortical necrosis.
* Seropositivity for Epstein-Barr virus (EBV)
* negative pregnancy test and agreement on the use of effective contraception throughout the study

Exclusion Criteria:

* Presence of Donor Specific Antibody during kidney transplant or appeared at 3 months post-transplantation.
* seropositivity for HIV
* another history of other solid organ transplants (outside the kidney)
* primary non-function (persistence of a need for dialysis at 3 months post-transplantation)
* participation in progress to another interventional clinical study
* any clinical condition that the investigator considers incompatible with the course of the study.
* contraindication to belatacept and Tacrolimus
* Pregnant or breastfeeding woman
* Inability of the patient to comply with study procedures
* Person placed under guardianship or curatorship, under safeguard of justice

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2027-05-03 (Estimated); Study Completion 2027-05-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a transient replacement of CNIs by belatacept in renal transplant patients with early graft dysfunction. Creatinine clearance did not decrease by more than 25% from the cessation of belatacept 6 months after reintroduction of CNI. | Month 15
  Feasibility was defined by preserved renal function and good tolerance 6 months after reintroduction of CNI.
  Renal function was defined as preserved if creatinine clearance (according to Chronic Kidney Disease - Epidemiology Collaboration (CKD-EPI)) did not decrease by more than 25% from the cessation of belatacept.
  The good tolerance of CNI was defined by the absence of complications leading to the cessation of treatment.

SECONDARY OUTCOMES:
Evaluate the effectiveness of belatacept treatment on renal function (creatinine clairance) and to prevent rejection. (Number of rejection épisodes) | Day 0, Month 3, Month 6, Month 9
  Longitudinal monitoring of renal function (Day 0, Month 3, Month 6, Month 9) and collection of rejection episodes.
Evaluate the tolerance of treatments (belatacept during phase 1 and CNI during phase 2). Number of adverse events. | Month 3, Month 6, Month 9, Month 12, Month 15
  Collection of infectious episodes and neoplasias
Estimate the cost of care (from 3 months to 18 months post-transplant) and compare with the cost of a theoretical arm benefiting from belatacept continuously and a theoretical arm benefiting from CNIs continuously. | Month 3, Month 6, Month 9, Month 12, Month 15
  Number of care resources used for treatment : number of medication, number of hospitalization, number of transportation, number of consultations, number of medical procedures, possible home help and associated costs over 15 months of follow-up, and collection of cost data in the literature for the comparison.
Evaluate the evolution of the quality of life during the 15 months of follow-up and compare it to a theoretical arm benefiting from belatacept continuously, and a theoretical arm benefiting from CNIs continuously: generic EuroQol-5D scale | Month 3, Month 6, Month 9, Month 12, Month 15
  Measurement of quality of life scores (generic EuroQol-5D scale) every 3 months for 15 months and collection of quality of life data in the literature for comparison.
Evaluate the differential impact of SNFs and belatacept on cell populations of the immune system | Month 3, Month 6, Month 9, Month 12, Month 15
  Differential analysis of cell populations by standardised flow cytometry combined with unbiased analysis.
Evaluate the differential impact of NICs and belatacept on the level of CMV replication and its clinical consequences. | Month 3, Month 6, Month 9, Month 12, Month 15
  Longitudinal monitoring of CMV PCR

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, Loire Atlantique, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Le Meur Y, Aulagnon F, Bertrand D, Heng AE, Lavaud S, Caillard S, Longuet H, Sberro-Soussan R, Doucet L, Grall A, Legendre C. Effect of an Early Switch to Belatacept Among Calcineurin Inhibitor-Intolerant Graft Recipients of Kidneys From Extended-Criteria Donors. Am J Transplant. 2016 Jul;16(7):2181-6. doi: 10.1111/ajt.13698. Epub 2016 Mar 2. PMID 26718625
- [Result] Vincenti F. Belatacept and Long-Term Outcomes in Kidney Transplantation. N Engl J Med. 2016 Jun 30;374(26):2600-1. doi: 10.1056/NEJMc1602859. No abstract available. PMID 27355541